CLINICAL TRIAL: NCT02181634
Title: A Multi-Institutional, Single Arm, Two-Stage Phase II Trial of Nab-Paclitaxel and Gemcitabine for First-Line Treatment of Patients With Advanced or Metastatic Cholangiocarcinoma
Brief Title: Phase II Trial of Nab-Paclitaxel and Gemcitabine for First-Line Treatment of Patients With Cholangiocarcinoma
Acronym: PrE0204
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PrECOG, LLC. (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PrE0204; AX-CL-OTHER-PrECOG-004080 (Other Grant/Funding Number: Celgene); 2015-002066-24 (EudraCT Number)
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Cholangiocarcinoma
Keywords: Advanced Cholangiocarcinoma; Metastatic Cholangiocarcinoma; CCA; Bile Duct Cancer; Nab-Paclitaxel; Abraxane®; Gemcitabine; Gemzar®
MeSH Terms: conditions — Cholangiocarcinoma; Bile Duct Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nab-Paclitaxel and Gemcitabine (Experimental): Nab-Paclitaxel 125 mg/m² IV and Gemcitabine 1000 mg/m² on days 1, 8 and 15 every 28 days until progression or unacceptable toxicity.
  Interventions: Drug: Nab-Paclitaxel and Gemcitabine

INTERVENTIONS:
Drug: Nab-Paclitaxel and Gemcitabine — Nab-Paclitaxel will be administered first, at a dose of 125 mg/m² IV over a period of 30 minutes; gemcitabine will be administered second, at a dose of 1000 mg/m² over a period of 30 minutes.
  Other Names: Abraxane®; Cytotoxic Antimicrotubular; Gemzar®; Pyrimidine Antimetabolite

SUMMARY:
Patients with advanced or metastatic cholangiocarcinoma (CCA) who are not eligible for curative surgery, transplantation, or ablative therapies will receive nab-paclitaxel and gemcitabine chemotherapy.

The purpose of this study is to evaluate the effectiveness and safety of the combination of nab-paclitaxel and gemcitabine. The effectiveness will be determined by improvement in the length of time during and after treatment, that the CCA does not get worse.

DETAILED DESCRIPTION:
Advanced cholangiocarcinomas (CCAs) are aggressive tumors with median survival time after diagnosis of less than 12 months, and five-year overall survival (OS) of ~5% with systemic chemotherapy. Currently available systemic therapies for CCA are largely ineffective, thus the rationale for the proposed research is to investigate targeted delivery of chemotherapy.

The goal of this study is to evaluate the efficacy of gemcitabine plus nab-paclitaxel in patients with advanced CCA. This is based on the premise that nab-paclitaxel binds to SPARC (secreted protein acidic and rich in cysteine) through its interaction with albumin, leading to an increase in intra-tumoral concentration of gemcitabine through decreased deoxycytidine deaminase (CDA) enzyme. We hope to improve on the OS of patients with advanced CCA through the use of the synergistic combination of nab-paclitaxel and gemcitabine to specifically target the SPARC protein in the peri-tumoral stroma. We aim to provide critical data to further develop pharmacologic strategies to target the desmoplastic stroma in order to increase chemotherapy responsiveness of CCAs.

We will also examine whether circulating tumor cell (CTC) levels with targeted gene expression analysis and stromal SPARC levels correlate with patient outcome and thus serve as prognostic biomarkers. We will evaluate the role of Human Equilibrative Nucleoside Transporter 1 (hENT1), CDA and tumor fibrosis as additional prognostic and predictive biomarkers in CCA. This clinical trial hopes to improve on the poor prognosis of patients with advanced CCA by establishing the activity of a platinum-free doublet, nab-paclitaxel plus gemcitabine that has shown clear clinical benefit in pancreatic cancer which has close biological parallels to CCA.

A maximum of 70 patients will be enrolled to attain 67 eligible/evaluable patients. Stage I will enroll 37 patients. If 21 or more patients are alive and progression-free at 6 months, the study will proceed to Stage II and an additional 33 patients will be enrolled.

Procurement of archived tissue, if available, from a previous diagnostic biopsy is mandatory for enrollment. If not available, this will not preclude participation in the trial, nor will additional biopsies be performed for research purposes only.

Optional blood samples will be requested.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically-confirmed diagnosis of cholangiocarcinoma Stage II, III, or IV CCA (intra-hepatic, extra-hepatic and perihilar) that is not eligible for curative resection, transplantation, or ablative therapies. Tumors of mixed histology are not allowed.
* Must have radiographically measurable disease in at least one site not previously treated with radiation, chemoembolization, radioembolization, or other local ablative procedures; a new area of tumor progression within or adjacent to a previously-treated lesion, if clearly measurable by a Radiologist, is acceptable.
* May have received prior radiation, chemoembolization, radioembolization, or other local ablative therapies, or hepatic resection if completed ≥ 4 weeks prior to registration AND if patient has recovered to ≤ grade 1 toxicity. NOTE: Measurable disease (as required above) must still be present.
* May have received prior radiation for bone or brain metastases if patient is now asymptomatic and has completed all radiation and steroid therapy (if applicable) ≥ 2 weeks prior to registration.
* Age ≥ 18 years.
* Child-Pugh score of A or B with ≤ 7 points.
* Eastern Cooperative Oncology Group performance status of 0-1.
* Willing to provide archived tissue, if available, from a previous diagnostic biopsy.
* Must be able to tolerate CT and/or MRI with contrast.
* Adequate organ function obtained ≤ 2 weeks prior to registration:

  * Absolute Neutrophil Count ≥ 1500/mm³
  * Hemoglobin ˃9.0 g/dL
  * Platelets ˃100,000/mm³
  * Serum Creatinine ≤ 1.5x Upper Limit Normal (ULN)
  * Creatinine Clearance ≥ 50 mL/min
  * Albumin ≥ 2.8 g/dL
  * Total Bilirubin ≤ 1.5 mg/dL or ≤ 1.5x ULN
  * Aspartate Aminotransaminase (AST)/Alanine Aminotransaminase (ALT) ≤ 2.5x ULN (≤ 5x ULN in patients with liver metastases)
  * International Normalized Ratio (INR) <1.5x the ULN [INR ≥ 1.5 is allowed if anticoagulation is used.]
* Women must not be pregnant or breastfeeding since nab-paclitaxel and/or gemcitabine may harm the fetus or child.
* Must not have received prior systemic cytotoxic chemotherapy or targeted therapy for this cancer.
* Must not be receiving treatment with other investigational agents.
* Must not have a pre-existing >grade 2 peripheral neuropathy.
* Must not be receiving immunosuppressive medications, including systemic corticosteroids, aside from the following exceptions: used for adrenal replacement, appetite stimulation, therapy for asthma, bronchitis exacerbation (≤ 2 weeks), anti-emesis, or pre-medication for procedures (i.e. CT scan).
* No known Hepatitis B, Hepatitis C, or Human Immunodeficiency Virus (HIV) seropositivity.
* Must not have undergone liver transplantation.
* Must not have serious non-healing wound, ulcer, bone fracture, or abscess.
* Must not have undergone a major surgical procedure <4 weeks prior to registration.
* Must not have possible histories of pneumonitis or pneumonitis risk factors.
* Must not have an active second malignancy other than non-melanoma skin cancer or cervical carcinoma in situ.
* Must have no ongoing or active, uncontrolled infections.
* Must have no evidence of significant, uncontrolled concomitant diseases including, but not limited to: symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, myocardial infarction within preceding 12 months, uncontrolled peripheral vascular disease, cerebrovascular accident within preceding 12 months, pulmonary disease impairing functional status or requiring oxygen, connective tissue disease including lupus.
* Must not have any history of allergic reaction(s) attributed to compounds of similar composition to nab-paclitaxel or gemcitabine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-12-09 (Actual); Primary Completion 2016-09-24 (Actual); Study Completion 2017-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vaibhav Sahai, MD, Study Chair — University of Michigan Health System in Ann Arbor, MI
Locations (25):
- United States (24):
  - Colorado Cancer Research Program, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - Ochsner Medical Center, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - University Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - St. Joseph Mercy Health System, Ann Arbor, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Metro Minnesota CCOP, Saint Louis Park, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Mount Sinai Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pennsylvania; Abramson Cancer Center at Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Gundersen Health System, La Crosse, Wisconsin
  - University of Wisconsin-Madison, Madison, Wisconsin
  - Aurora Cancer Care, Wauwatosa, Wisconsin
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Data is proprietary

REFERENCES:
- [Result] Sahai V, Catalano PJ, Zalupski MM, Lubner SJ, Menge MR, Nimeiri HS, Munshi HG, Benson AB 3rd, O'Dwyer PJ. Nab-Paclitaxel and Gemcitabine as First-line Treatment of Advanced or Metastatic Cholangiocarcinoma: A Phase 2 Clinical Trial. JAMA Oncol. 2018 Dec 1;4(12):1707-1712. doi: 10.1001/jamaoncol.2018.3277. PMID 30178032

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nab-Paclitaxel and Gemcitabine
Started | 74
Eligible and Treated | 73
Completed | 2
Not Completed | 72
Not completed — Lack of Efficacy | 33
Not completed — Adverse Event | 17
Not completed — Physician Decision | 8
Not completed — Withdrawal by Subject | 5
Not completed — Death | 2
Not completed — Treatment delayed greater than 4 weeks | 3
Not completed — Ineligible | 1
Not completed — Max number of dose reduction | 1
Not completed — Symptomatic progression | 1
Not completed — Patient opted to proceed to surgery | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Nab-Paclitaxel and Gemcitabine
Number analyzed (Participants) | 73
Age, Continuous [Median (Full Range); unit: years] | 62 [36 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 71
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 67
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Rate at 6 Months (Proportion of Participants Alive and Progression-Free at 6 Months)
Description: Progression-free survival is defined as the time from the date of first study treatment to either the date of documented disease progression or death from any cause, whichever occurred first. Progression-free survival rate at 6 months is defined as the proportion of patients who were disease progression-free and alive at 6 months.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the diameter/axes of target lesions, taking as reference the smallest sum on study, or unequivocal progression of existing non-target lesions, or the appearance of new lesions.
Time Frame: Assessed at 6 months
Population: Eligible and treated
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Nab-Paclitaxel and Gemcitabine
Number analyzed (Participants) | 73
proportion of participants | 0.605 [0.482 to 0.729]

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from enrollment until death or last patient contact.
Time Frame: Every 3-6 months for up to 3 years
Population: Eligible and treated
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel and Gemcitabine
Number analyzed (Participants) | 73
months | 11.2 [9.6 to 14.7]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the time from the date of first study treatment to either the date of documented disease progression or death from any cause, whichever occurred first.
Time Frame: Every 3-6 months for up to 3 years
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel and Gemcitabine
Number analyzed (Participants) | 73
months | 7.7 [5.9 to 13.1]

4. Secondary Outcome: Time To Progression (TTP)
Description: TTP was defined as the time from date of first dose of study therapy to date of removal from study for progression. Patients who have not experienced progression were censored at the date of last disease evaluation. Progression is evaluated using Solid Tumor Response Criteria (RECIST) Version 1.1. Progression is defined as at least a 20% increase in the sum of the diameters/axes of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm over the nadir. The appearance of new lesions or unequivocal progression of existing non-target lesions also constitutes disease progression.
Time Frame: Every 3-6 months for up to 3 years
Population: Eligible and treated
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel and Gemcitabine
Number analyzed (Participants) | 73
months | 7.7 [6.5 to 13.1]

5. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate is defined as the proportion of patients with complete response or partial response per RECIST version 1.1. Complete response is defined as disappearance of all lesions. Partial response is defined as at least a 30% decrease in the sum of the diameters/axes of target lesions and the persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker levels above the normal limits. A confirmation assessment performed >=4 weeks after the criteria for response is met is required.
Time Frame: Every 3-6 months for up to 3 years
Population: Eligible and treated
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Nab-Paclitaxel and Gemcitabine
Number analyzed (Participants) | 73
proportion of participants | 0.301 [0.199 to 0.420]

6. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate is the proportion of patients achieved complete response, partial response or stable disease per RECIST version 1.1. Complete response is defined as disappearance of all lesions. Partial response is defined as at least a 30% decrease in the sum of the diameters/axes of target lesions and the persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker levels above the normal limits. Stable disease is defined as neither sufficient shrinkage to qualify for complete or partial response nor sufficient increase to qualify for progression. A confirmation assessment performed >=4 weeks after the criteria for response is met is required.
Time Frame: Every 3-6 months for up to 3 years
Population: Eligible and treated patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Nab-Paclitaxel and Gemcitabine
Number analyzed (Participants) | 73
proportion of participants | 0.658 [0.537 to 0.765]

7. Secondary Outcome: Association Between PFS and Maximum Change in Carbohydrate Antigen (CA) 19-9 From Baseline
Description: Patients were dichotomized into maximum CA 19-9 decline >=50% and maximum CA 19-9 decline <50%. Cox proportional hazards model was used to evaluate the association between PFS and maximum change in CA 19-9.
Time Frame: CA 19-9 was evaluated every 8 weeks until progression or for up to 3 years and off-treatment
Population: Eligible and treated patients with CA 19-9 data available
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel and Gemcitabine
Number analyzed (Participants) | 35
months
  CA 19-9 decline >=50%: number analyzed (Participants) | 26
  CA 19-9 decline >=50% | 7.7 [6.6 to 13.1]
  CA 19-9 decline <50%: number analyzed (Participants) | 9
  CA 19-9 decline <50% | 1.9 [1.6 to 18.2]
Statistical Analysis 1: Comparison: Nab-Paclitaxel and Gemcitabine; Test type: Superiority; p = 0.099, Log Rank; Hazard Ratio (HR) = 2.02, 95% CI 2-sided [0.86 to 4.75]

8. Secondary Outcome: Association Between OS and Maximum Change in Carbohydrate Antigen (CA) 19-9 From Baseline
Description: Patients were dichotomized into maximum CA 19-9 decline >=50% and maximum CA 19-9 decline <50%. Cox proportional hazards model was used to evaluate the association between OS and maximum change in CA 19-9.
Time Frame: CA 19-9 was evaluated every 8 weeks until progression or for up to 3 years and off-treatment
Population: Eligible and treated patients with CA 19-9 data available
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel and Gemcitabine
Number analyzed (Participants) | 35
months
  CA 19-9 decline >=50%: number analyzed (Participants) | 26
  CA 19-9 decline >=50% | 14.6 [10.2 to 25.6]
  CA 19-9 decline <50%: number analyzed (Participants) | 9
  CA 19-9 decline <50% | 10.2 [4.1 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.
Statistical Analysis 1: Comparison: Nab-Paclitaxel and Gemcitabine; Test type: Superiority; p = 0.34, Log Rank; Hazard Ratio (HR) = 1.54, 95% CI 2-sided [0.64 to 3.71]

9. Other Pre Specified Outcome: Change in Circulating Tumor Cells (CTCs)
Description: Correlate change in CTCs to median PFS, OS, TTP, ORR and DCR.
Time Frame: Prior to Cycle 1, Day 1; Cycle 1 Day 8; Cycle 3, Day 1 and at Off Treatment
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Stromal SPARC Expression
Description: Correlate stromal SPARC (high versus low) expression by immunohistochemistry (IHC) with median PFS, OS, TTP, ORR and DCR.
Time Frame: Baseline
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Fibrosis Expression
Description: Correlate fibrosis (low, intermediate and high) by trichrome staining with median PFS, OS, TTP, ORR and DCR.
Time Frame: Baseline
Reporting Status: Not Posted

12. Other Pre Specified Outcome: CDA Expression
Description: Correlate CDA (high versus low) expression by IHC with median PFS, OS, TTP, ORR and DCR.
Time Frame: Baseline
Reporting Status: Not Posted

13. Other Pre Specified Outcome: hENT Expression
Description: Correlate hENT1 (high versus low) expression by IHC with median PFS, OS, TTP, ORR and DCR.
Time Frame: Baseline
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Banking Biospecimens for Future Assessment
Description: Optional specimen banking of patient blood specimens (including serum, plasma and buffy coat) as well as fixed left-over tissue specimens when available from all enrolled patients in this trial for possible future molecular, pharmacogenomic, and/or proteomic testing.
Time Frame: Prior to Cycle 1, Day 1; Cycle 1, Day 8; Cycle 3, Day 1 and at Off Treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every week for the first 2 cycles, then every two cycles (every 8 weeks) and 30 days after the last dose of therapy
Arm/Group | Nab-Paclitaxel and Gemcitabine
Serious Adverse Events (participants affected / at risk) | 42/74
Other Adverse Events (participants affected / at risk) | 72/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Paclitaxel and Gemcitabine (N=74)
Anemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 2
Fatigue (General disorders) | 1
Generalised oedema (General disorders) | 2
Multi-organ failure (General disorders) | 2
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 5
Bile duct obstruction (Hepatobiliary disorders) | 1
Bile duct stenosis (Hepatobiliary disorders) | 2
Biliary fistula (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 3
Cholecystitis (Hepatobiliary disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 3
Abscess (Infections and infestations) | 1
Biliary tract infection (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 1
Emphysematous cholecystitis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 4
Humerus fracture (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 3
Embolism (Vascular disorders) | 3
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Paclitaxel and Gemcitabine (N=74)
Abdominal distension (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 12
Acute kidney injury (Renal and urinary disorders) | 5
Alanine aminotransferase increased (Investigations) | 18
Alopecia (Skin and subcutaneous tissue disorders) | 39
Anemia (Blood and lymphatic system disorders) | 31
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Ascites (Gastrointestinal disorders) | 5
Aspartate aminotransferase increased (Investigations) | 18
Asthenia (General disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6
Blood alkaline phosphatase increased (Investigations) | 17
Blood bilirubin increased (Investigations) | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Chills (General disorders) | 11
Constipation (Gastrointestinal disorders) | 34
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Decreased appetite (Gastrointestinal disorders) | 28
Deep vein thrombosis (Vascular disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 7
Diarrhea (Gastrointestinal disorders) | 35
Dizziness (Nervous system disorders) | 11
Dry mouth (Gastrointestinal disorders) | 4
Dysgeusia (Nervous system disorders) | 17
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 22
Embolism (Vascular disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11
Fatigue (General disorders) | 53
Headache (Nervous system disorders) | 6
Hot flashes (Vascular disorders) | 6
Hyperbilirubinemia (Investigations) | 7
Hypertension (Vascular disorders) | 10
Hypoalbuminemia (Investigations) | 9
Hypocalcemia (Investigations) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 8
Influenza like illness (General disorders) | 4
Insomnia (Psychiatric disorders) | 12
Leukopenia (Investigations) | 5
Mucosal inflammation (Infections and infestations) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 14
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Nail discolouration (Skin and subcutaneous tissue disorders) | 5
Nausea (Gastrointestinal disorders) | 34
Neuropathy peripheral (Nervous system disorders) | 28
Neutropenia (Blood and lymphatic system disorders) | 26
Neutrophil count decreased (Investigations) | 14
Oedema peripheral (General disorders) | 31
Pain (General disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Peripheral sensory neuropathy (Nervous system disorders) | 9
Platelet count decreased (Investigations) | 11
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5
Pyrexia (General disorders) | 18
Rash (Skin and subcutaneous tissue disorders) | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Sepsis (Infections and infestations) | 4
Stomatitis (Gastrointestinal disorders) | 8
Thrombocytopenia (Investigations) | 16
Tremor (Nervous system disorders) | 4
Vision blurred (Eye disorders) | 5
Vomiting (Gastrointestinal disorders) | 18
Weight decreased (Investigations) | 22
Weight increased (Investigations) | 5
White blood cell count decreased (Investigations) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No